CLINICAL TRIAL: NCT03449823
Title: Are Renal Artery Doppler Indices Different Between Monochorionic Diamniotic Twins With Twin-twin Transfusion Syndrome and Monochorionic Diamniotic Twins Without Twin-twin Transfusion Syndrome?
Brief Title: Renal Artery Dopplers in Twin Twin Transfusion Syndrome
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Russell Miller, Assistant Professor of Obstetrics and Gynecology, Columbia University
Other Study IDs: AAAQ9660
Record Dates: First submitted 2018-02-07; First posted 2018-02-28 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Twin Twin Transfusion Syndrome
Keywords: Renal Artery Doppler
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TTTS Cases: Cases of monochorionic / diamniotic twin pregnancies diagnosed with twin-twin transfusion syndrome.
  Interventions: Diagnostic Test: Doppler ultrasound of fetal renal artery
- MCDA Controls: Controls of monochorionic / diamniotic twin pregnancies without a diagnosis of twin-twin transfusion syndrome.
  Interventions: Diagnostic Test: Doppler ultrasound of fetal renal artery

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound of fetal renal artery — Doppler ultrasound assessment of the proximal fetal renal artery to with measurement of the peak systolic velocity, resistive index, pulsatility index, and systolic/diastolic ratio.

SUMMARY:
Twin-twin transfusion syndrome (TTTS) is a complication affecting 10-15% of monochorionic, diamniotic (MCDA) twin pregnancies. Unevenly distributed blood flow across a shared placental circulation results in a volume-restricted donor twin and a volume-overloaded recipient twin, and TTTS has high perinatal morbidity and mortality without treatment.

Differential donor and recipient findings in TTTS can be observed upon ultrasound evaluation. TTTS is classified according to the Quintero staging system, which evaluates amniotic fluid volumes, fetal bladders, Doppler study of the umbilical artery and ductus venosus, and for the presence of hydrops or death. However, due to seemingly complex and variable disease pathophysiology, the Quintero system cannot predict outcomes on a case-by-case basis.

Prior studies have associated fetal renal artery Doppler ultrasound measurements with amniotic fluid volume in singleton pregnancies. In fetuses with placental insufficiency, adaptive circulatory changes maintain adequate oxygen delivery to vital organs such as the heart, brain, and adrenals, with a consequent deprivation to splanchnic organs. In the fetal kidney, as vascular resistance increases during hypoxia, renal perfusion decreases proportionately. These changes are reflected in renal artery Doppler findings. As these same adaptations are believed to occur in donor twins, renal artery Doppler studies may also be of value in the TTTS evaluation.

This study plans to perform renal artery Doppler assessments in MCDA twins complicated by TTTS, and compare them to measurements in gestational-age equivalent MCDA twins without TTTS. If findings differ significantly, it would support further investigation into the use of renal artery Doppler studies for the evaluation of complicated MCDA twins.

DETAILED DESCRIPTION:
TTTS, which complicates 10-15% of MCDA twin pregnancies, is characterized by a net imbalance of volume between twins, mediated through abnormal placental blood vessel anastomoses that connect the two placental circulations. Clinically, the "donor" twin develops features of anemia and hypovolemia, while the "recipient" twin shows signs of hypervolemia and hypertensive fluid overload. If untreated, the syndrome has a perinatal mortality rate as high as 80-100%. Although modern intrauterine therapies have improved the rates of fetal death, significant risks of morbidity and mortality remain even after treatment.

Twin-twin transfusion syndrome is most commonly classified according to a staging system developed by Quintero et al in 1999, which is based on discrete, categorical ultrasound findings (amniotic fluid volume, presence/absence of a fetal bladder, umbilical artery Doppler studies, fetal hydrops, and death). The system includes 5 stages ranging from mild disease with isolated discordant amniotic fluid volumes, to severe disease with demise of one or both twins. Although this system has some prognostic value, it also has significant limitations due to the highly complex physiologic conditions that are involved in the disease. For example, some criteria in the staging system are not consistently representative of fetal physiology. Additionally, the stages do not correlate well with overall perinatal survival or with outcomes following intrauterine therapies.

Recent work has demonstrated that the complex pathophysiology of twin-twin transfusion syndrome involves a discordant activation of the renin angiotensin system (RAS). RAS is normally important in fluid and salt regulation in both the adult and the fetus, and TTTS in marked hypovolemia and hypervolemia in monozygous fetuses within the same maternal environment. The renal RAS in the donor is up-regulated, presumably as a consequence of hypovolemia. The recipient is also exposed to high levels or RAS components, either due to the transfusion of these components from the donor via anastomoses, or via discordant placental RAS activation, resulting in a hypertensive, hypervolemic state.

Multiple studies have identified a correlation between Doppler assessment of the fetal renal artery and the development of oligohydramnios, a hypovolemic state, in singleton pregnancies. However, the use of renal artery Doppler studies has not yet been fully evaluated in twin gestations. In particular, it has not been evaluated in MCDA twin gestations complicated by TTTS, the pathophysiology of which involves significant alterations in fetal volume and fluid status.

This project is intended to serve as a single-center study to determine if there is indeed a difference in renal artery Doppler parameters in sets of MCDA twins with TTTS compared to sets of MCDA twins without TTTS. The identification of a significant difference would potentially provide support for further investigation into this measurement as a screening tool or prognostic indicator when applied to MCDA twin pregnancies.

Secondary goals of this study include: comparing donor to recipient renal artery Doppler findings among pregnancies with TTTS, evaluating serial renal artery Doppler findings over time per pregnancy, and evaluating pre- and post-therapy renal artery Doppler findings in those pregnancies undergoing therapy for TTTS.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with monochorionic / diamniotic (MCDA) twin pregnancies with and without twin-twin transfusion syndrome (TTTS)
* greater than 14 weeks gestation

Exclusion Criteria:

* higher-order multiple gestation
* sonographic evidence of a major structural fetal anomaly (exceptions to this structural fetal anomaly exclusion are acquired recipient twin cardiac changes that are known to be associated with TTTS - these cases may be considered for study inclusion)

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The subject population will consist of pregnant women with monochorionic / diamniotic (MCDA) twin pregnancies with and without twin-twin transfusion syndrome (TTTS). This population is selected in order to investigate twin-twin transfusion syndrome, which is a disease process that is unique to pregnancies with monochorionic / diamniotic twins. Patients will be included in the study if they have a diagnosis of a MCDA twin gestation beyond the first trimester or pregnancy (greater than 14 weeks gestation).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Fetal renal artery Doppler PSV for twin A | Obtained at the time of enrollment.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the peak systolic velocity for twin A.
Fetal renal artery Doppler RI for twin A | Obtained at the time of enrollment.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the resistive index for twin A.
Fetal renal artery Doppler PI for twin A | Obtained at the time of enrollment.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the pulsatility index for twin A.
Fetal renal artery Doppler PSV for twin B | Obtained at the time of enrollment.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the peak systolic velocity for twin B.
Fetal renal artery Doppler RI for twin B | Obtained at the time of enrollment.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the resistive index for twin B.
Fetal renal artery Doppler PI for twin B | Obtained at the time of enrollment.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the pulsatility index for twin B.

SECONDARY OUTCOMES:
Post-laser fetal renal artery Doppler PSV for twin A | Obtained within one week following fetoscopic laser therapy for cases in which this treatment is provided.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the peak systolic velocity for twin A.
Post-laser fetal renal artery Doppler RI for twin A | Obtained within one week following fetoscopic laser therapy for cases in which this treatment is provided.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the resistive index for twin A.
Post-laser fetal renal artery Doppler PI for twin A | Obtained within one week following fetoscopic laser therapy for cases in which this treatment is provided.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the pulsatility index for twin A.
Post-laser fetal renal artery Doppler PSV for twin B | Obtained within one week following fetoscopic laser therapy for cases in which this treatment is provided.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the peak systolic velocity for twin B.
Post-laser fetal renal artery Doppler RI for twin B | Obtained within one week following fetoscopic laser therapy for cases in which this treatment is provided.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the resistive index for twin B.
Post-laser fetal renal artery Doppler PI for twin B | Obtained within one week following fetoscopic laser therapy for cases in which this treatment is provided.
  Doppler ultrasound assessment of the proximal fetal renal artery with measurement of the pulsatility index for twin B.

CONTACTS AND LOCATIONS:
Overall Officials: Joses Jain, MD, Study Director — Columbia University; Russell Miller, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Society for Maternal-Fetal Medicine; Simpson LL. Twin-twin transfusion syndrome. Am J Obstet Gynecol. 2013 Jan;208(1):3-18. doi: 10.1016/j.ajog.2012.10.880. Epub 2012 Nov 27. PMID 23200164
- [Background] Lewi L, Jani J, Blickstein I, Huber A, Gucciardo L, Van Mieghem T, Done E, Boes AS, Hecher K, Gratacos E, Lewi P, Deprest J. The outcome of monochorionic diamniotic twin gestations in the era of invasive fetal therapy: a prospective cohort study. Am J Obstet Gynecol. 2008 Nov;199(5):514.e1-8. doi: 10.1016/j.ajog.2008.03.050. Epub 2008 Jun 4. PMID 18533114
- [Background] Acosta-Rojas R, Becker J, Munoz-Abellana B, Ruiz C, Carreras E, Gratacos E; Catalunya and Balears Monochorionic Network. Twin chorionicity and the risk of adverse perinatal outcome. Int J Gynaecol Obstet. 2007 Feb;96(2):98-102. doi: 10.1016/j.ijgo.2006.11.002. Epub 2007 Jan 23. PMID 17250837
- [Background] Fusi L, Gordon H. Twin pregnancy complicated by single intrauterine death. Problems and outcome with conservative management. Br J Obstet Gynaecol. 1990 Jun;97(6):511-6. doi: 10.1111/j.1471-0528.1990.tb02521.x. PMID 2198920
- [Background] van Heteren CF, Nijhuis JG, Semmekrot BA, Mulders LG, van den Berg PP. Risk for surviving twin after fetal death of co-twin in twin-twin transfusion syndrome. Obstet Gynecol. 1998 Aug;92(2):215-9. doi: 10.1016/s0029-7844(98)00159-8. PMID 9699754
- [Background] Ong SS, Zamora J, Khan KS, Kilby MD. Prognosis for the co-twin following single-twin death: a systematic review. BJOG. 2006 Sep;113(9):992-8. doi: 10.1111/j.1471-0528.2006.01027.x. Epub 2006 Aug 10. PMID 16903844
- [Background] Quintero RA, Morales WJ, Allen MH, Bornick PW, Johnson PK, Kruger M. Staging of twin-twin transfusion syndrome. J Perinatol. 1999 Dec;19(8 Pt 1):550-5. doi: 10.1038/sj.jp.7200292. PMID 10645517
- [Background] Taylor MJ, Govender L, Jolly M, Wee L, Fisk NM. Validation of the Quintero staging system for twin-twin transfusion syndrome. Obstet Gynecol. 2002 Dec;100(6):1257-65. doi: 10.1016/s0029-7844(02)02392-x. PMID 12468171
- [Background] Yamamoto M, El Murr L, Robyr R, Leleu F, Takahashi Y, Ville Y. Incidence and impact of perioperative complications in 175 fetoscopy-guided laser coagulations of chorionic plate anastomoses in fetofetal transfusion syndrome before 26 weeks of gestation. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 2):1110-6. doi: 10.1016/j.ajog.2005.07.003. PMID 16157121
- [Background] Taylor GM, Peart WS, Porter KA, Zondek LH, Zondek T. Concentration and molecular forms of active and inactive renin in human fetal kidney, amniotic fluid and adrenal gland: evidence for renin-angiotensin system hyperactivity in 2nd trimester of pregnancy. J Hypertens. 1986 Feb;4(1):121-9. doi: 10.1097/00004872-198602000-00019. PMID 3007602
- [Background] Galea P, Barigye O, Wee L, Jain V, Sullivan M, Fisk NM. The placenta contributes to activation of the renin angiotensin system in twin-twin transfusion syndrome. Placenta. 2008 Aug;29(8):734-42. doi: 10.1016/j.placenta.2008.04.010. Epub 2008 Jun 16. PMID 18558429
- [Background] Arduini D, Rizzo G. Fetal renal artery velocity waveforms and amniotic fluid volume in growth-retarded and post-term fetuses. Obstet Gynecol. 1991 Mar;77(3):370-3. PMID 1992401
- [Background] Stigter RH, Mulder EJ, Bruinse HW, Visser GH. Doppler studies on the fetal renal artery in the severely growth-restricted fetus. Ultrasound Obstet Gynecol. 2001 Aug;18(2):141-5. doi: 10.1046/j.1469-0705.2001.00493.x. PMID 11529994
- [Background] Oz AU, Holub B, Mendilcioglu I, Mari G, Bahado-Singh RO. Renal artery Doppler investigation of the etiology of oligohydramnios in postterm pregnancy. Obstet Gynecol. 2002 Oct;100(4):715-8. doi: 10.1016/s0029-7844(02)02203-2. PMID 12383539
- [Background] Azpurua H, Dulay AT, Buhimschi IA, Bahtiyar MO, Funai E, Abdel-Razeq SS, Luo G, Bhandari V, Copel JA, Buhimschi CS. Fetal renal artery impedance as assessed by Doppler ultrasound in pregnancies complicated by intraamniotic inflammation and preterm birth. Am J Obstet Gynecol. 2009 Feb;200(2):203.e1-11. doi: 10.1016/j.ajog.2008.11.001. PMID 19185102
- [Background] Benzer N, Pekin AT, Yilmaz SA, Kerimoglu OS, Dogan NU, Celik C. Predictive value of second and third trimester fetal renal artery Doppler indices in idiopathic oligohydramnios and polyhydramnios in low-risk pregnancies: a longitudinal study. J Obstet Gynaecol Res. 2015 Apr;41(4):523-8. doi: 10.1111/jog.12601. Epub 2014 Nov 3. PMID 25363086